CLINICAL TRIAL: NCT00779480
Title: Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Study of KW-2449 in Acute Myelogenous Leukemia
Brief Title: Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Study of KW-2449 in Acute Myelogenous Leukemia (AML) (Protocol Number: 2449-US-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Failure to demonstrate a tolerable dose that had potential for efficacy.
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2449-US-002
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Acute Myelogenous Leukemia (AML)
Keywords: Acute Myelogenous Leukemia; Safety; Dose Tolerance; Pharmacokinetics/Pharmacodynamics; FLT-3
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — KW 2449

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KW-2449 (Experimental): Sequential dose escalation in separate cohorts of 3+3 design from 450 mg/day to 800 mg/day total daily dose.
  Interventions: Drug: KW-2449

INTERVENTIONS:
Drug: KW-2449 — KW-2449 50 mg capsules administered 3 or 4 times per day for 21-day cycles up to 6 cycles

SUMMARY:
To determine the maximum tolerated dose of KW-2449 in people with acute myelogenous leukemia who are not candidates for approved therapy. As well, the study will determine the response rate to KW-2449.

DETAILED DESCRIPTION:
Phase 1: To determine the maximum tolerated daily dose (MTDD) of KW 2449 when administered to subjects with AML who are not candidates for approved therapy.

This was originally a Phase 1/Phase 2 study. However, a tolerable dose that had the potential for efficacy could not be identified in Phase 1. Therefore, Phase 2 was never conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of AML (excluding acute promyelocytic leukemia) that has relapsed or was not responsive to prior chemotherapy.

   Phase 2: Only subjects with the FLT3/ITD mutation will be enrolled in Phase 2.
2. Eastern Cooperative Oncology Group (ECOG) Scale score17 of 0, 1, or 2 (refer to Appendix 1);
3. Male or female, at least 18 years of age;
4. Signed written informed consent;
5. Serum creatinine ≤ 2.0 mg/dL;
6. Serum SGOT (AST) and SGPT (ALT) ≤ 5x the upper limits of normal (ULN); serum bilirubin ≤ 2 mg/dL (serum bilirubin must be ≤ 3.0 mg/dL in any subject with Gilbert's Syndrome); and
7. For women of childbearing potential, a negative serum pregnancy test must be obtained prior to administration of KW-2449.

Exclusion Criteria:

1. Subjects who are candidates for approved therapies for their underlying condition;
2. Prior treatment with KW-2449;
3. Concomitant treatment with chemotherapy (systemic or intrathecal), radiotherapy, immunotherapy, or any investigational agent;
4. Evidence of active central nervous system (CNS) leukemia;
5. Previous or concurrent malignancy except noninvasive non-melanomatous skin cancer, in situ carcinoma of the cervix, or other solid tumor treated curatively, and without evidence of recurrence for at least 2 years prior to study entry;
6. Uncontrolled systemic infection (viral, bacterial, or fungal);
7. Uncontrolled disseminated intravascular coagulopathy;
8. Major surgery within the 28 days preceding the first dose KW-2449;
9. Radiotherapy within the 28 days preceding the first dose KW-2449, or lack of recovery from any radiotherapy-related acute adverse event;
10. Treatment with approved systemic therapy for the underlying hematologic condition within 14 days of the first dose of KW-2449 with the exception of hydroxyurea (Hydrea®) or leukapheresis for hyperleukocytosis and/or thrombocytosis (see Concomitant Medication and Treatment), or lack of recovery from any adverse event from prior systemic therapy.
11. Treatment with another investigational agent within the 28 days preceding the first dose of KW-2449, or lack of recovery from any adverse event from such treatment;
12. Known positive serology for human immunodeficiency virus (type 1 and/or 2);
13. Clinically significant cardiac dysfunction (New York Heart Association Class 3 or 4) at the time of screening, or a history of myocardial infarction or heart failure within 3 months preceding the first dose of KW-2449;
14. Chronic Graft versus Host Disease (GVHD) with the exception of mild (Grade 1) skin GVHD;
15. Phase 1 only: ≥ Grade 2 nausea or vomiting within 7 days preceding the first dose KW 2449;
16. Active autoimmune disease requiring immunosuppressive therapy;
17. Female subjects who are pregnant or breast feeding; Pregnant women are excluded from this study because the embryotoxic potential of KW-2449 is unknown. It is not known whether KW-2449 passes into human breast milk. Nursing mothers should not use KW-2449.
18. Male or female subjects of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with the institution's standards; Pregnancy should be avoided in women receiving KW 2449 and in female partners of men receiving KW-2449. All subjects receiving KW-2449 should implement appropriate contraceptive methods.
19. Known current drug or alcohol abuse;
20. Other severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may compromise the safety of the subject during the study, affect the subject's ability to complete the study, or interfere with interpretation of study results;
21. Subject is judged by the Investigator to be inappropriate for study participation for any reason, including an inability to communicate or cooperate with the Investigator;
22. Use of hematopoietic growth factors (i.e., such as erythropoietin or darbepoetin alfa, filgrastim [granulocyte colony-stimulating factor {G-CSF}], sargramostim [granulocyte-macrophage colony-stimulating factor {GM-CSF}], or thrombopoietic agents) within 14 days preceding the first dose of KW-2449; or
23. Monoamine oxidase-B (MAO-B) or aldehyde oxidase (AOX) inhibitors within 7 days preceding the first dose KW-2449.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety as determine by adverse event rate and dose limiting toxicity | Approximately 6 months

SECONDARY OUTCOMES:
Hematologic activity/improvement, Pharmacokinetics/Pharmacodynamics | Approximately 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - St. Francis Hospital, Greenville, South Carolina

REFERENCES:
- [Background] Pratz KW, Cortes J, Roboz GJ, Rao N, Arowojolu O, Stine A, Shiotsu Y, Shudo A, Akinaga S, Small D, Karp JE, Levis M. A pharmacodynamic study of the FLT3 inhibitor KW-2449 yields insight into the basis for clinical response. Blood. 2009 Apr 23;113(17):3938-46. doi: 10.1182/blood-2008-09-177030. Epub 2008 Nov 24. PMID 19029442
- [Background] Shiotsu Y, Kiyoi H, Ishikawa Y, Tanizaki R, Shimizu M, Umehara H, Ishii K, Mori Y, Ozeki K, Minami Y, Abe A, Maeda H, Akiyama T, Kanda Y, Sato Y, Akinaga S, Naoe T. KW-2449, a novel multikinase inhibitor, suppresses the growth of leukemia cells with FLT3 mutations or T315I-mutated BCR/ABL translocation. Blood. 2009 Aug 20;114(8):1607-17. doi: 10.1182/blood-2009-01-199307. Epub 2009 Jun 18. PMID 19541823